CLINICAL TRIAL: NCT04172714
Title: Theragnostic Low Dose Y90 Microspheres for Personalized Y90 Radioembolization Dosimetry Planning
Brief Title: Low-dose Y90 Treatment Planning for HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nima Kokabi, Assistant professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00112192
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Results first posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: HCC; Cancer of Liver; Cancer
Keywords: Cancer; Radiation therapy; Liver Diseases; Radiology, Interventional; Radiology
MeSH Terms: conditions — Liver Neoplasms; Neoplasms; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Second mapping with low-dose Y90 (Experimental): Patients will undergo standard of care mapping study with 99TC-MAA to plan for Y90 radioembolization therapy. Additionally,non-standard of care, intervention will be to do a second mapping study using SIR-spheres microspheres with low-dose Y90 (15 mCi) before the therapeutic Y90 radioembolization.
  Interventions: Device: SIR-Spheres microspheres

INTERVENTIONS:
Device: SIR-Spheres microspheres — SIR-Spheres® Y-90 resin microspheres consist of biocompatible polymer resin microspheres of a median diameter of 32.5 microns (range between 20 and 60 microns) loaded with yttrium-90 (beta radiation penetrating an average of 2.5 mm in tissue to destroy tumor cells). The resin microspheres are small enough to become lodged in the arterioles within the growing rim of the tumor but are too large to pass through the capillaries and into the venous system. Since yttrium-90 has a half-life of 64.1 hours, most of the radiation (94%) is delivered to the tumor over 11 days.
  Other Names: SIRSPHERE; Y90 resin-based microspheres

SUMMARY:
The study proposes low-dose Y90 microspheres for therapy planning of HCC, as an alternative to Technetium (99mTc) albumin aggregated (MAA), to be a bioidentical therapeutic Y90 surrogate marker to better predict and thus achieve optimal therapeutic dosing.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is a second deadliest cancer in the world with less than 20% of patients eligible for curative surgery at the time of diagnosis. Yttrium-90 (Y90) radioembolization is palliative treatment with promising result. However, one of the most important factors in the success of Y90 treatment is to ensure adequate dose of radioactive material is delivered to the tumor. The technetium-99 macroaggregated albumin (MAA) which is currently used for Y90 treatment planning and shunt study does not predict distribution of Y90 in the lungs, tumors, and liver. Therefore, accurate and personalized treatment planning cannot be performed using MAA. In this study, we are proposing using low-dose Y90 microspheres for the planning stage of the therapy to obtain an accurate estimation of distribution of Y90 therapy dose. This will in turn allow us to ensure adequate dose of Y90 is delivered to the tumor(s) while minimizing dose delivered to non-tumor liver and lungs in order to decrease the chance of treatment related toxicity to the liver and lungs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years
2. Life expectancy of 6 months or more as determined by the investigator
3. HCC confirmed by Liver Reporting & Data System (LIRADS) on MRI or CT
4. Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) with CT scan, MRI, or calipers by clinical exam. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
5. ≤3 lesions
6. Longest dimension of the largest lesion ≤7cm
7. Single lobe disease
8. No significant extrahepatic metastatic disease
9. Barcelona Clinic Liver Cancer Stage A, B or C
10. ECOG < 2 (Appendix A)
11. Lesion(s) <50% of liver volume
12. Bilirubin ≤ 2 mg/dL
13. Albumin ≥ 3 g/dL
14. PT/INR < 2
15. AST/ALT ≤ 3 institutional upper limit of normal (ULN)
16. Platelet count > 50,000/mcL
17. Lung shunt fraction of <20% by planar MAA if dose modification results in inadequate dose delivered to the tumor(s)
18. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
19. Completion of all previous therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥ 12 week before the start of study therapy. Willingness and ability of the subject to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions.

u. Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation. v. The effects of Y90 microspheres on the developing human fetus are unknown. For this reason female of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy. Winship Protocol #: RAD4784 Version Date: Aug 22, 2019 20 | P a g e w. FCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of [IND Agent] administration. A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months

Exclusion Criteria:

* An individual who does not meet all the inclusion criteria in section.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nima Kokabi, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kokabi N, Webster LA, Dabbous H, Shah A, Brandon D, Galt J, Xing M, Villalobos A, Davarpanahfakhr A, Kappadath SC, Schuster DM. Resin-Based 90 Y Tumor Dose as a Predictor of Duration of Response and Survival in Patients With Surgically Unresectable Hepatocellular Carcinoma : A Prospective Single-Arm Study. Clin Nucl Med. 2024 Sep 1;49(9):799-805. doi: 10.1097/RLU.0000000000005198. Epub 2024 May 21. PMID 38861361
- [Derived] Kokabi N, Arndt-Webster L, Chen B, Brandon D, Sethi I, Davarpanahfakhr A, Galt J, Elsayed M, Bercu Z, Cristescu M, Kappadath SC, Schuster DM. Voxel-based dosimetry predicting treatment response and related toxicity in HCC patients treated with resin-based Y90 radioembolization: a prospective, single-arm study. Eur J Nucl Med Mol Imaging. 2023 May;50(6):1743-1752. doi: 10.1007/s00259-023-06111-9. Epub 2023 Jan 18. PMID 36650357
- [Derived] Kokabi N, Webster LA, Elsayed M, Switchenko JM, Chen B, Brandon D, Galt J, Sethi I, Cristescu M, Kappadath SC, Schuster DM. Accuracy and Safety of Scout Dose Resin Yttrium-90 Microspheres for Radioembolization Therapy Treatment Planning: A Prospective Single-Arm Clinical Trial. J Vasc Interv Radiol. 2022 Dec;33(12):1578-1587.e5. doi: 10.1016/j.jvir.2022.08.027. Epub 2022 Sep 6. PMID 36075560

RESULTS

PARTICIPANT FLOW:
Groups:
- Technetium-99m Macroaggregated Albumin (99mTc-MAA)/Second Mapping With Low-dose Y90: Patients will undergo standard of care mapping study with 99TC-MAA to plan for Y90 radioembolization therapy. Additionally,non-standard of care, intervention will be to do a second mapping study using SIR-spheres microspheres with low-dose Y90 (15 mCi) before the therapeutic Y90 radioembolization.
  Additionally, non-standard of care, intervention will be to do a second mapping study using SIR-Spheres microspheres: SIR-Spheres® Y-90 resin microspheres consist of biocompatible polymer resin microspheres of a median diameter of 32.5 microns (range between 20 and 60 microns) loaded with yttrium-90 (beta radiation penetrating an average of 2.5 mm in tissue to destroy tumor cells). The resin microspheres are small enough to become lodged in the arterioles within the growing rim of the tumor but are too large to pass through the capillaries and into the venous system. Since yttrium-90 has a half-life of 64.1 hours, most of the radiation (94%) is delivered to the tumor over 11 days.
Period: Overall Study
Arm/Group | Technetium-99m Macroaggregated Albumin (99mTc-MAA)/Second Mapping With Low-dose Y90
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Technetium-99m Macroaggregated Albumin (99mTc-MAA)/ Second Mapping With Low-dose Y90: Patients will undergo standard of care mapping study with 99TC-MAA to plan for Y90 radioembolization therapy. Following MAA, non-standard of care, intervention will be to do a second mapping study using SIR-spheres microspheres with low-dose Y90 (15 mCi) before the therapeutic Y90 radioembolization.
  SIR-Spheres microspheres: SIR-Spheres® Y-90 resin microspheres consist of biocompatible polymer resin microspheres of a median diameter of 32.5 microns (range between 20 and 60 microns) loaded with yttrium-90 (beta radiation penetrating an average of 2.5 mm in tissue to destroy tumor cells). The resin microspheres are small enough to become lodged in the arterioles within the growing rim of the tumor but are too large to pass through the capillaries and into the venous system. Since yttrium-90 has a half-life of 64.1 hours, most of the radiation (94%) is delivered to the tumor over 11 days.
Arm/Group | Technetium-99m Macroaggregated Albumin (99mTc-MAA)/ Second Mapping With Low-dose Y90
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Lung Shunt Fraction (LSF) Ratio
Description: Y-90 radioembolization treatment requires estimating the activity shunted from the liver to the lungs, referred to as a lung shunt fraction (LSF). It is expressed in ratios, with higher ratio meaning a higher transit of Y-90 to the lungs (worse outcome) and lower ratio, lower transit of Y-90 to the lungs (better outcome).
Time Frame: Baseline
Population: Participants underwent standard of care and then underwent second mapping with low dose Y90 intervention.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Technetium-99m Macroaggregated Albumin (99mTc-MAA): All patients will undergo standard of care mapping study with Technetium-99m macroaggregated albumin (99mTc-MAA) to plan for Y90 radioembolization therapy.
Arm/Group | Technetium-99m Macroaggregated Albumin (99mTc-MAA) | Second Mapping With Low-dose Y90
Number analyzed (Participants) | 30 | 30
Ratio | 5.68 (3.12) | 5.79 (2.08)

2. Primary Outcome: Tumor to Normal Liver Activity Ratio (TNR)
Description: The ratios of the tumor-to-normal liver parenchymal radioactivity uptake count will be measured. TNR values will be calculated by dividing the mean count of the tumorous volume of interest (VOI) by the mean count of normal liver.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Technetium-99m Macroaggregated Albumin (99mTc-MAA) | Second Mapping With Low-dose Y90
Number analyzed (Participants) | 30 | 30
Ratio | 2.67 (1.67) | 2.75 (1.2)

3. Secondary Outcome: Number of Participants With Tumor Response Using Imaging Modified Response Criteria in Solid Tumors (m-RECIST) Post Y90 Embolization
Description: To identify tumor dose response threshold (TDRT) using Imaging Modified Response Criteria in Solid Tumors (m-RECIST), that is a method for measuring treatment response and measure of antitumor activity of cytotoxic drugs. This is measured using imaging: CT or MRI. The overall response is a combination of responses in each category: complete response (disappearance of any intramural arterial enhancement in all target lesions), partial response (at least 30% decrease in the sum of the diameters of viable target lesions), stable disease (any cases that do not qualify for either partial response or progressive disease) or progressive disease (an increase of at least 20% in the sum of the diameters of viable, enhancing target lesions, taking as a reference the smallest sum of the diameters of viable target lesions recorded since treatment started).
Time Frame: 6 months post intervention
Measure: Number; unit: Count of participants
Arm/Group | Technetium-99m Macroaggregated Albumin (99mTc-MAA)/ Second Mapping With Low-dose Y90
Number analyzed (Participants) | 30
Count of participants
  Complete tumor response | 23
  Partial tumor response | 3
  Stable disease | 6
  Progression of disease | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: All subjects underwent standard of care mapping study with 99TC-MAA to, immediately followed by a non-standard of care intervention: Second mapping study using SIR-spheres microspheres with low-dose Y90 for radioembolization. Both interventions were done on the same day and one immediately after the other. All data for adverse events was collected following all interventions, up to 6 months after the interventions, hence there is no distinction among arms for adverse events.
Arm/Group | Technetium-99m Macroaggregated Albumin (99mTc-MAA)/Second Mapping With Low-dose Y90
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Technetium-99m Macroaggregated Albumin (99mTc-MAA)/Second Mapping With Low-dose Y90 (N=30)
Transplantation complication (Hepatobiliary disorders) | 1 (30)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Technetium-99m Macroaggregated Albumin (99mTc-MAA)/Second Mapping With Low-dose Y90 (N=30)
Fatigue (General disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Elevated Bilirubin (Blood and lymphatic system disorders) | 5 (5)
Elevated ALT (Blood and lymphatic system disorders) | 11 (11)
Elevated AST (Blood and lymphatic system disorders) | 11 (11)
Decreased Albumin (Blood and lymphatic system disorders) | 2 (2)
Elevated Creatinine (Blood and lymphatic system disorders) | 2 (2)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Decreased WBC count (Blood and lymphatic system disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Altered platelet count (Blood and lymphatic system disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT04172714/Prot_SAP_003.pdf
  • Informed Consent Form (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT04172714/ICF_004.pdf